CLINICAL TRIAL: NCT02362698
Title: Clinical Research of Electro-acupuncture Combined Psychological Intervention on Internet Addiction Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-07LQ04
Record Dates: First submitted 2015-01-03; First posted 2015-02-13 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Addiction
MeSH Terms: conditions — Behavior, Addictive | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- electro-acupuncture (Experimental): Receiving electro-acupuncture treatment once every other day, half an hour per treatment, 10 times as one treatment course, subjects received 2 courses of treatment.
  Interventions: Other: electro-acupuncture
- psychological intervention (Active Comparator): Receiving cognitive behavioral therapy once every four days, each time two hours. Five times intervention as one treatment course, subjects received 2 courses of treatment.
  Interventions: Other: psychological intervention

INTERVENTIONS:
Other: electro-acupuncture — 13points were selected including he-gu(LI4), nei-guan(PC6), tai-chong(LR3) and san-yin-jiao(SP6) from both sides, bai-hui(GV20) and si-shen-cong(EX-HN1) from head.
  HANS-200A acupoints stimulator, which had two output channels, was connected to some selected points. Dilatational wave was adopted in this research, the frequency of rarefaction wave was 2 hertz and condensation wave was 100 hertz, with a waviness width of 0.3ms. Switched the stimulator on after connected the poles to the needles, adjusted the intensity of output gradually from 0 milliampere to the extent of subject's maximum tolerance. Then needles would be remained on the body for half an hour.
  Arms: electro-acupuncture
Other: psychological intervention — Cognitive behavioral therapy was adopted by national accredited professional psychologist, in the form of team work and individual counseling, aim to help IA participants to understand their deviant behaviors, correct unhealthy cognitive states and eventually retrieve normal life style.
  Arms: psychological intervention

SUMMARY:
this research adopted multicentered, randomly and parallel control methods to observe the clinical effects of electro-acupuncture combined psychological intervention on internet addiction disorder, aim to provide a convenient, affordable and effective clinical protocol.

DETAILED DESCRIPTION:
This research was aimed to discuss the impact of acupuncture treatment on the impulsive behavior of Internet Addiction Disorder (IAD) sufferers, with the detection of magnetic resonance spectroscopy (MRS), the assessment of Young's Internet Addiction Test (IAT), Barratt Impulsivity Scale (BIS-11) and Go/No-go task, hopefully that this research could provide basis for the further study as well as the establishment of comprehensive assessment and treatment protocol of IAD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects manifested three or more among the seven following conditions within one year could be defined as internet addiction:
* (1) Tolerance, complied with either one: ①Satisfaction obtaining through markedly increasing time online ②Spending same period of time online but with dramatic declining satisfaction.
* (2) Any following symptoms appeared after quitting internet surfing: ①Obvious withdrawal syndrome: A-- Quitted or decreased long time internet surfing. B--Within one month after A, two or more following symptoms appeared: (a) Depressed. (b) Psychomotor fidgety. (c) Compulsively thought things happened online. (d) Hallucinated or dreamed about internet related stuff. (e) Consciously or unconsciously carried out tapping the keyboard movement. C--The symptoms in B led to unexpected damage to one's social life, work and other important aspects of life, even depression. ②Desperate to surf the internet or seek similar online service in a bid to relieve or avoid withdrawal syndrome.
* (3) More frequent online behaviors or longer online time than planned.
* (4) Had been trying hard to reduce or control internet use but never succeeded.
* (5) Spent large amount of time on internet related things, such as purchasing online books, trying out new browsers, organizing downloaded files, etc.
* (6) Giving up or reducing important social, work or entertainment activities.
* (7) Despite unfavorable physical, mental, social or work consequences, continued to use internet.

Exclusion Criteria:

* Other psychiatric disease history.
* Drug addiction history
* Severe cardiovascular disease, blood diseases, malignant tumors or any other contraindication of electro-acupuncture.
* Allergic to acupuncture treatment.
* Participants with intracranial diseases or abnormal scalp structure.
* Participants with metal implant.
* Color blindness, left handedness.
* Women in gestation or lactation period.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
the change of the level of brain N-acetylaspartate on magnetic resonance spectroscopy from baseline at 40 days | day 1 and the day after treatment(treatment covered 40 days) had completed
  analysis
the change from baseline of the total scores on Internet Addiction Test(IAT) at 40 days | day 1 and the day after treatment(treatment covered 40 days) had completed
  questionnaire
the change of the level of brain choline on magnetic resonance spectroscopy from baseline at 40 days | day 1 and the day after treatment(treatment covered 40 days) had completed
  analysis

CONTACTS AND LOCATIONS:
Overall Officials: Tianmin Zhu, Doctor, Study Chair — Chengdu University of Traditional Chinese Medicine

REFERENCES:
- [Derived] Peng W, Wang Y, Hao Q, Wang J, Chen Y, Qiu M, Tu Y, Li H, Zhu T. Effects of Electroacupuncture Combined With Psychological Intervention on Depressive Status and Contingent Negative Variation in Patients With Internet Addiction Disorder: A Randomized Controlled Trial. Front Psychiatry. 2021 Nov 15;12:722422. doi: 10.3389/fpsyt.2021.722422. eCollection 2021. PMID 34867514